CLINICAL TRIAL: NCT05946369
Title: Preoperative Neutrophils to Lymphocytes Ratio in Predicting the Response to BCG in Non-muscle Invasive Bladder Cancer
Brief Title: Neutrophils to Lymphocytes Ratio in Predicting the Response to BCG in Non-muscle Invasive Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, principle investigator, Ain Shams University
Other Study IDs: MS 475/ 2021
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Urinary Bladder Cancer; Urinary Bladder Neoplasm; BCG; Trans Urethral Resection of a Bladder Tumor; Non-Muscle Invasive Bladder Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neutrophil to lymphocyte ratio less than 3: Patients are classified into 2 groups according to NLR < or ≥ 3 and follow up the 2 groups for recurrence or regression of bladder urothelial tumor and documentation of BCG failure
  Interventions: Diagnostic Test: Neutrophil to lymphocyte ratio
- Neutrophil to lymphocyte ration more than or equal 3: Patients are classified into 2 groups according to NLR < or ≥ 3 and follow up the 2 groups for recurrence or regression of bladder urothelial tumor and documentation of BCG failure
  Interventions: Diagnostic Test: Neutrophil to lymphocyte ratio

INTERVENTIONS:
Diagnostic Test: Neutrophil to lymphocyte ratio — Complete blood count with differential to evaluate the Neutrophil to lymphocyte ratio for each patient

SUMMARY:
There is a relation between inflammatory cells and the prognosis of tumors (cancer colon, renal, liver, and urinary bladder).

In this study, the investigators will link the Neutrophils to Lymphocytes ratio to the response to intravesical BCG therapy post trans-urethral resection of urinary bladder tumors for the non-invasive urinary bladder tumors.

DETAILED DESCRIPTION:
The gold standard treatment for non-invasive urinary bladder tumors is by transurethral resection of bladder tumor (TURBT) and a re-TURBT when indicated, followed by adjuvant intravesical immunotherapy (BCG). However, the recurrence and progression rates of non-muscle invasive bladder cancer (NMIBC) for 5 years range from 31% to 78% and from 1% to 45%, respectively.

To improve personalized care, prognostic models have been developed to help in prediction of the high-risk patients and recurrence helping in clinical and therapeutic decision-making. These models are based on standard clinic-pathological features such as T stage, grade, multifocality, sex, tumor diameter, recurrence rate, and concomitant carcinoma in situ.

According to the current theories, the systemic inflammatory response triggered by cancer leads to relative neutrophilia and lymphocytopenia, creating a pro-oncogenic inflammatory condition. An elevated NLR (Neutrophil to lymphocyte ratio) implies that cell-mediated immunity is impaired and systemic inflammation is increased in inflammatory processes. Among patients with non-invasive urinary bladder tumors, an elevated NLR (Neutrophil to lymphocyte ratio) was described in the literature to be associated with advanced pathologic stage, invasiveness, and bad prognosis.

The study aims to assess the role of preoperative Neutrophils to Lymphocytes ratio as a predictor for the response to BCG in patients with non-muscle invasive bladder cancer in patients following trans-urethral resection of bladder tumor (TURBT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-muscle invasive urothelial tumor of the urinary bladder

Exclusion Criteria:

1. Concomitant malignancy.
2. Hematological disorders.
3. History of radiation or chemotherapy.
4. Concomitant infection or chronic inflammatory diseases.
5. Missing preoperative differential blood cell count.
6. Patients with low grade non muscle invasive Urinary baldder tumors.
7. Patients missing BCG after biopsy revealing NMIBC.
8. patients with non-compliance to BCG doses or the scheduled follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with intermediate and high-risk group of non-muscle invasive urothelial tumor will be included in our study.
  They will go through detailed history taking, general and local examinations. Routine Labs (specially CBC with Differential Count) preoperatively will be done to all patients during the surgery workup.
  Histopathology report of the first resection and another one of the check cystoscopy to confirm the primary diagnosis.
  BCG course ( once weekly for 6 weeks) 2-6 weeks after resection as an induction course. Then maintaince doses for 1-3 years based on the European Association of Urology recommendations.
  Follow up cystoscopy will be scheduled based on the European association of Urology schedule for intermediate and high risk groups.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
BCG failure | 3 years following tumor resection and BCG instillation
  evaluation of tumor recurrence or progression post BCG intravesical instillation in our study population and draw up and correlation between BCG failure and Neutrophil to lymphocyte ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No